

## **School of Sport, Exercise and Health Sciences**

## Influence of High-fat Overfeeding on Circulating Hepatokine Concentrations: A Randomised Crossover Study

17<sup>th</sup> November 2017

## **OVEREAT Study Statistical Analysis Plan**

The data collected will be analysed using the software package SPSS (SPSS Version 23, SPSS Inc., Chicago, IL) and an alpha value of P < 0.05 will be set to indicate statistical significance. Parametric assumptions will be checked using the Shapiro-Wilk test in order to confirm normal distribution of the data. Two-hour area under the curve (AUC) calculations for plasma glucose and insulin during the oral glucose tolerance tests will be performed using the trapezoidal method. Whole-body insulin sensitivity will be calculated using the Matsuda Insulin Sensitivity Index (ISI) equation:

$$\frac{10,000}{\sqrt{(Glucose_{0\,min}\times Insulin_{0\,min}\times mean\,Glucose_{OGTT}\times mean\,Insulin_{OGTT})}}$$

The homeostatic model assessment of insulin resistance (HOMA-IR) will also be calculated using the formula:

$$\frac{Glucose_{0 min} \times Insulin_{0 min}}{22.5}$$

Adipose tissue insulin resistance (ADIPO-IR) will be calculated using the formula:

$$Insulin_{0 min} \times NEFA_{0 min}$$

A one-way repeated measures analysis of variance (ANOVA) will be performed to assess differences in daily energy intake, daily fat intake and 7-day physical activity and sedentary behaviour (i.e sitting time, standing time, light physical activity, moderate-vigorous physical activity) between the high-fat condition, control condition and baseline measurement.

For the outcome measures which will be taken only pre- and post-dietary conditions, a 2 x 2 repeated measures ANOVA will be used for analysis. This includes the following outcome measures: Body fat percentage, resting metabolic rate, fat oxidation percentage, glucose AUC, insulin AUC and Matsuda ISI.

For the outcome measures which will be taken both pre-diet and post-diet as well as one and three days into the diet, a 2 x 4 repeated measures ANOVA will be used for analysis. This includes fasting plasma concentrations of: LECT2, FGF21, fetuin-A, acylated ghrelin, PYY, CTX, P1MP, glucose, insulin, NEFA and triglycerides. These outcome measures also include: HOMA-IR, ADIPO-IR, subjective ratings of appetite, food preference, body mass and both systolic and diastolic blood pressure.

Where a significant interaction effect is observed, *post hoc* paired samples *t*-tests with a Bonferroni correction will be used to locate any differences. If Mauchly's test of sphericity is violated by any variables, Greenhouse-Geisser corrected values will be used.